CLINICAL TRIAL: NCT03575676
Title: Phase IIa, Double-blind, Randomized, Placebo-controlled Study of the Efficacy and Safety of SOM3355 in Huntington's Disease (HD) Patients With Chorea Movements.
Brief Title: Efficacy and Safety of SOM3355 in Huntington's Disease Chorea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOM Innovation Biotech SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOMCT02; 2018-000203-16 (EudraCT Number)
Record Dates: First submitted 2018-06-11; First posted 2018-07-02 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Huntington's Chorea
Keywords: Huntington; Chorea; SOM3355
MeSH Terms: conditions — Huntington Disease; Chorea | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Administration of SOM3355 100mg BID for 6 weeks, SOM3355 200mg BID for 6 weeks, SOM3355 100mg BID for 6 weeks and placebo BID for 6 weeks.
  Interventions: Drug: SOM3355 100mg BID; Drug: SOM3355 200mg BID; Drug: Placebo BID
- Group B (Experimental): Administration of placebo BID for 6 weeks, SOM3355 100mg BID for 6 weeks, SOM3355 200mg BID for 6 weeks and SOM3355 100mg BID for 6 weeks.
  Interventions: Drug: SOM3355 100mg BID; Drug: SOM3355 200mg BID; Drug: Placebo BID

INTERVENTIONS:
Drug: SOM3355 100mg BID — Oral
Drug: SOM3355 200mg BID — Oral
Drug: Placebo BID — Oral

SUMMARY:
Phase IIa study to evaluate the efficacy and safety of SOM3355 in chorea movements associated with Huntington's disease

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age at time of consent.
* Diagnosis of HD definite by a movement disorders expert and confirmed by a number of HTT gene CAG repeats equal or greater than 36.
* Female of child bearing potential (FCBP) and non-vasectomized male agree to practice appropriate methods of birth control.
* Ability to walk independently or with minimal assistance.
* UHDRS TMC score equal or greater than 8.
* UHDRS TFC equal or greater than 4.
* Subject has provided written informed consent or through his/her legally authorized representative.

Exclusion Criteria:

* Onset of HD symptoms prior to age 18 (Juvenile forms of HD).
* Non-ambulatory patients.
* A past medical history of clinically significant ECG abnormalities or a family history (grandparents, parents and siblings) of a prolonged QT-interval syndrome.
* Pregnant or breastfeeding female patients, including those planning to conceive during the period of the trial.
* Patients with psychiatric symptoms, or other impairments, that would interfere with their full compliance with the Investigator instructions and testing, unless there is an identified caregiver to support the patient.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study. The Investigator should make this determination in consideration of the subject's medical history and/or clinical laboratory test results at screening and baseline.
* Known allergy/sensitivity/intolerance to the study drugs or their excipients.
* Any significant laboratory results which, in the Investigator's opinion, would not be compatible with study participation or represent a risk for the subject while in the study.
* Prescribed anti-hypertensive medication, tetrabenazine, deutetrabenazine or valbenazine within 15 days prior starting the investigational treatment.
* Excluded concomitant medications: any anti-hypertensive medication, tetrabenazine, deutetrabenazine or valbenazine, all typical neuroleptics and all MAO inhibitors
* Subject has a history of alcohol or substance abuse in the previous 12 months.
* Patients with diabetic ketoacidosis or metabolic acidosis.
* Patients with cardiogenic shock, congestive heart failure, pulmonary hypertension due to right-sided heart failure, severe sinus bradycardia, atrioventricular block (grades II and III) or sinoatrial block.
* Subject has participated in an investigational drug or device trial within 30 days prior starting the investigational treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
UHDRS (Unified Huntington's Disease Rating Scale) Total Maximal Chorea (TMC) score | 6 months
  UHDRS subscore used to measure the effectiveness of SOM3355 on HD chorea.

SECONDARY OUTCOMES:
Clinical Global Impression of Change (CGIC) scale | 6 months
  PGIC reflects clinician's belief about the efficacy of treatment.
Patient Global Impression of Change (PGIC) scale | 6 months
  PGIC reflects a patient's belief about the efficacy of treatment.
UHDRS Total Functional Capacity (TFC) | 6 months
  A standardized rating scale used to assess capacity to work, handle finances, perform domestic chores and self-care tasks.
UHDRS Functional Assessment | 6 months
  Functional Assessment should be judged according to the investigator's opinion of capacity to perform the activity rather than the actual performance of this activity.
UHDRS Gait score | 6 months
  UHDRS subscore used to assess patient's gait.
UHDRS Total Motor Score (TMS) | 6 months
  Categoric clinical rating scale assessing multiple domains of motor disability in HD.
Columbia Suicide Severity Rating Scale (C-SSRS) | 6 months
  International validated questionnaire used for suicide assessment.
Safety (number of participants with adverse events) | 6 months
  The maximum grade for each type of AE will be recorded for each subject, and frequency tables will be presented and reviewed to determine patterns. The relationship of the AE to the study treatment will be taken into consideration. Hypotension and cardiovascular events will be specifically analyzed.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat

REFERENCES:
- [Derived] Gamez J, Calopa M, Munoz E, Ferre A, Huertas O, McAllister K, Reig N, Scart-Gres C, Insa R, Kulisevsky J. A proof-of-concept study with SOM3355 (bevantolol hydrochloride) for reducing chorea in Huntington's disease. Br J Clin Pharmacol. 2023 May;89(5):1656-1664. doi: 10.1111/bcp.15635. Epub 2022 Dec 28. PMID 36494329
- See also: SOM Biotech website — http://www.sombiotech.com